CLINICAL TRIAL: NCT02518425
Title: Which Instrumental Acoustic Voice Parameters Indicate Vocal Improvement After Voice Therapy in Patients With Functional Dysphonia
Brief Title: Improvement in Acoustic Voice Characteristics in Functional Dysphonia After Therapy
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BJ_02_02_2015
Record Dates: First submitted 2015-04-09; First posted 2015-08-07 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Functional Voice Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In a retrospective analysis of already existing clinical assessment data from patients with functional voice disorders the following aspects will be sampled, encoded and analysed: Outcomes pre and post treatment of

1. subjective voice symptoms measured by Voice Handicap Index (VHI-9i),
2. perceptual voice symptoms according to Grading-Roughness-Breathiness-Asthenia-Strain Scale (GRBAS Scale),
3. instrumental acoustic analysis parameters Jitter (%), speaking voice profile: mean and range of speaking pitch and intensity, max. intensity and mean pitch of calling voice, singing voice: min./max. and range of pitch and intensity, maximum phonation time, Dysphonia Severity Index (DSI).

ELIGIBILITY:
Inclusion Criteria:

* informed consent; patients 20 to 70 years with functional voice disorder; -diagnostics and voice therapy at University Hospital Zurich;
* full pre- and post treatment voice assessment (videostroboscopy, subjective self- assessment, instrumental acoustic and perceptual analysis).

Exclusion Criteria:

* known neurologic and psychiatric disease,
* hearing disorder,
* surgery of the head and neck area or intubation (for any reason) in last 18 months.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with functional voice disorders
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Instrumental acoustic voice parameters | Before (initial diagnosis) and after voice therapy, expected average of 11-20 weeks after initial diagnosis)
  Instrumental acoustic parameters are determined by a computer-assisted analysis of voice recordings. In the present study the following parameters are measured before and after voice therapy: Jitter % (deviation of fundamental frequency), mean and range of speaking pitch and intensity, maximum intensity and mean pitch of calling voice, minimum and max. and range of pitch and intensity of the singing voice, and the composite measure Dysphonia Severity Index (DSI).

SECONDARY OUTCOMES:
Subjective voice symptoms | Before (initial diagnosis) and after voice therapy, expected average of 11-20 weeks after initial diagnosis)
  Subjective voice symptoms are measured before and after voice therapy by the patient questionnaire "Voice Handicap Index" (VHI-9i).
Perceptual voice symptoms | Before (initial diagnosis) and after voice therapy, expected average of 11-20 weeks after initial diagnosis)
  Perceptual (hearable) voice symptoms are determined by the examiner before and after voice therapy using GRBAS Scale (Grading-Roughness-Breathiness-Asthenia-Strain Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Joerg E Bohlender, MD, Principal Investigator — University Hospital Zurich, Department of Otorhinolaryngology
Locations (1):
- Clinic for Otorhinolaryngology University Hospital Zurich, Zurich, Canton of Zurich, Switzerland